CLINICAL TRIAL: NCT06211088
Title: Famotidine Versus Placebo in Emergency Pediatric Surgery As a Risk to Postoperative Nausea and Vomiting ꞉ a Comparative Study by Gastric Ultrasound Measurement
Brief Title: Famotidine Versus Placebo in Emergency Pediatric Surgery As a Risk to Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Zaher Zaki Zaher, Director, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Aswu/721/1/23
Record Dates: First submitted 2023-12-26; First posted 2024-01-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nausea,vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- famotidine plus10ml normal saline (Active Comparator): Group A:(n. 25) will receive a 5 mg of famotidine that will be diluted to 10ml normal saline in 2 minutes preinduction.
  Interventions: Drug: famotidine plus10ml normal saline
- 10ml normal saline (Placebo Comparator): Group B: Controlled group (n. 25) will receive a10ml normal saline preinduction.
  Interventions: Other: 10ml normal saline

INTERVENTIONS:
Drug: famotidine plus10ml normal saline — to evaluate the difference of the gastric volume by quantitative measurements of gastric antrum preoperatively and postoperatively by using 5mg famotidine
  Arms: famotidine plus10ml normal saline
Other: 10ml normal saline — to evaluate the difference of the gastric volume by quantitative measurements of gastric antrum preoperatively and postoperatively by placebo
  Arms: 10ml normal saline

SUMMARY:
The aim of this study is to evaluate the difference of the gastric volume by quantitative measurements of gastric antrum preoperatively and postoperatively by using 5mg famotidine versus placebo as a risk factor of PONV.

DETAILED DESCRIPTION:
Gastric ultrasound examinations will be performed preoperatively and postoperatively on patients undergoing emergency surgery in pediatric. Gastric cross-sectional area (CSA) will be measured, in order to estimate the gastric volume. The data that will be obtained will be used to evaluate a difference of the gastric volume between the two groups preoperatively and postoperatively and the possible relationship between the gastric volume difference and postoperative adverse event (PONV).

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics patients aging between 2-13 years .
* pediatrics undergo urgent surgery (i.e., surgery that cannot be postponed for more than 48 h since clinical onset).
* PatientPediatrics come in trauma

Exclusion Criteria:

* PatientPediatrics severly shocked .
* PatientPediatrics with diffusely distended abdomen as this will obstacle gastric ultrasound .
* PatientPediatrics with history of hypersenstivity to famotidine .
* PatientPediatrics with hepatic or renal impairments

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
to evaluate the difference of the gastric volume by quantitative measurements of gastric antrum by gastric ultrasound preoperatively and postoperatively by using 5mg famotidine versus placebo as a risk factor of postoperative nausea and vomiting | 12 months
  to evaluate the difference of the gastric volume by quantitative measurements of gastric antrum by gastric ultrasound preoperatively and postoperatively by using 5mg famotidine versus placebo as a risk factor of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Zaher, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No